CLINICAL TRIAL: NCT07406971
Title: Safety of Transmucosal Capsaicin for Chemical Sphenopalatine Ganglion Stimulation in Acute Ischemic Stroke Within 24 Hours of Symptom Onset: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Safety of Transmucosal Capsaicin Sphenopalatine Ganglion Stimulation in Acute Ischemic Stroke: A Randomized Placebo-Controlled Trial (Cap-SPGAS)
Acronym: Cap-SPGAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Centenario Hospital Miguel Hidalgo (Other)
Responsible Party: Principal Investigator, Juan Manuel Marquez Romero, Principal investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cap-SPGAS
Record Dates: First submitted 2026-02-06; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ischemic Stroke
Keywords: Acute ischemic stroke; Capsaicin; Sphenopalatine ganglion stimulation
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transmucosal Capsaicin (Experimental)
  Interventions: Drug: Capsaicin Transmucosal Oral Film
- Placebo Oral Film (Placebo Comparator)
  Interventions: Drug: Placebo Transmucosal Oral Film

INTERVENTIONS:
Drug: Capsaicin Transmucosal Oral Film — A dissolvable transmucosal oral film containing a low dose of capsaicin designed for local administration in the oral cavity. The formulation is intended to provide controlled mucosal exposure to capsaicin for investigational neuromodulatory stimulation of trigeminal-parasympathetic pathways potentially involved in cerebral blood flow regulation. The film is administered once under clinical supervision in addition to standard medical care for acute ischemic stroke.
  Arms: Transmucosal Capsaicin
Drug: Placebo Transmucosal Oral Film — A dissolvable transmucosal oral film identical in appearance, texture, and administration method to the active study film but without capsaicin. The placebo film is administered once under clinical supervision in addition to standard medical care for acute ischemic stroke to maintain blinding.
  Arms: Placebo Oral Film

SUMMARY:
This study will evaluate the safety and tolerability of a dissolvable oral film containing a very small dose of capsaicin (the compound that produces the "hot" sensation in chili peppers) in adults with acute ischemic stroke. The film is designed to stimulate nerves in the mouth that may activate the sphenopalatine ganglion, a structure involved in regulating blood flow to the brain. The main purpose of this study is to determine whether the capsaicin film can be given safely to patients with acute ischemic stroke when started within 24 hours of symptom onset.

Participants will be randomly assigned (like flipping a coin) to receive either the capsaicin oral film or a placebo film that looks and tastes similar but contains no capsaicin. Neither the participants nor the clinical team will know which film is given (double-blind). All participants will continue to receive standard medical care for acute ischemic stroke.

After administration of the study film, participants will be closely monitored for side effects and changes in vital signs (blood pressure, heart rate, respiratory rate, temperature, and oxygen saturation) at prespecified time points up to 72 hours. The primary outcome is the frequency of adverse events related to the study product within 72 hours after treatment begins. Participants will also be followed clinically up to 3 months as part of usual stroke care.

The results of this study will help determine whether this approach is safe and feasible, and whether further studies are warranted.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 80 years.

National Institutes of Health Stroke Scale (NIHSS) score between 6 and 20 at screening.

Symptom onset within 24 hours prior to study intervention.

Pre-stroke modified Rankin Scale (mRS) score ≤1.

Provision of written informed consent by the participant or legally authorized representative.

Exclusion Criteria:

Intracranial hemorrhage on neuroimaging.

Severe impairment of consciousness judged by the investigator to preclude safe participation.

Persistent blood pressure >220/120 mmHg after initial medical management.

Severe systemic disease that, in the investigator's judgment, may interfere with study participation or safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events Within 72 Hours After Administration | 72 hours after study intervention administration
  The primary outcome is the proportion of participants experiencing any adverse event within 72 hours after administration of the study oral film. Adverse events include any unfavorable clinical sign, symptom, or change in vital signs temporally associated with study treatment, regardless of causality. Vital signs (blood pressure, heart rate, respiratory rate, temperature, and oxygen saturation) are recorded at predefined time points during the first 72 hours.

SECONDARY OUTCOMES:
Change in Systolic Blood Pressure Over 72 Hours | Baseline (pre-dose) through 72 hours post-dose
  Change in systolic blood pressure (mmHg) from baseline (pre-dose) to each prespecified post-dose assessment time point through 72 hours. Values will be summarized by treatment group.
Change in Heart Rate Over 72 Hours | Baseline (pre-dose) through 72 hours post-dose
  Change in heart rate (beats per minute) from baseline (pre-dose) to each prespecified post-dose assessment time point through 72 hours. Values will be summarized by treatment group.
Treatment Tolerability Within 72 Hours | Up to 72 hours post-dose
  Proportion of participants who complete the assigned study oral film administration without discontinuation due to intolerance, and incidence of local tolerability symptoms (e.g., oral burning/irritation, excessive salivation, cough) within 72 hours after administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Centenario Hospital Miguel Hidalgo, Aguascalientes, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data underlying the results reported in publications may be shared with qualified researchers upon reasonable request, subject to institutional approval, data use agreements, and applicable privacy regulations.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning after publication of the primary study results and continuing for up to 5 years thereafter.
Access Criteria: Requests should include a methodologically sound proposal. Data sharing will require approval by the study investigators and execution of a data use agreement.

REFERENCES:
- [Background] Marquez-Romero JM, Huerta-Franco MR, Vargas-Luna M, Madrigal-Gutierrez CA, Esparza-Hernandez JM, Velazquez-Barcena MG. Dose Escalation and Safety of Capsaicin for Cerebral Perfusion Augmentation: A Pilot Study. Stroke. 2021 Jul;52(7):2203-2209. doi: 10.1161/STROKEAHA.120.032773. Epub 2021 May 10. PMID 33966493
- [Background] Marquez-Romero JM, Garcia-Perales C, Garcia-Arellano M, Ortiz MS, Perez-Malagon CD, Huerta-Franco MR, Vargas-Luna FM. Capsaicin for Cerebral Perfusion Augmentation: A Randomized Open-Label Trial. Stroke. 2024 Apr;55(4):e112-e114. doi: 10.1161/STROKEAHA.123.046045. Epub 2024 Mar 8. No abstract available. PMID 38456262